CLINICAL TRIAL: NCT04564118
Title: A Retrospective Analysis of the Adherence to Clinical Practice Guidelines Using the "MedicBK" Digital Platform in Patients With Hypertension and Atrial Fibrillation (the INTELLECT Trial)
Brief Title: A Retrospective Analysis of the Adherence to Clinical Practice Guidelines Using the "MedicBK" Digital Platform in Patients With Hypertension and Atrial Fibrillation
Acronym: INTELLECT
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Collaborators: Medicbook LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 909-2020
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Arterial Hypertension
Keywords: atrial fibrillation; arterial hypertension; digital medicine; Clinical Decision Support System
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: retrospective data on treatment from EMC
  Interventions: Drug: Retrospective analysis of assigned treatment
- Group 2: Treatment assignment using medicBC CDSS platform in the same cohort of patients

INTERVENTIONS:
Drug: Retrospective analysis of assigned treatment — analysis of treatment assigned by physicians within routine clinical practice
  Groups: Group 1

SUMMARY:
The Clinical Decision Support Systems (CDSS) based on real clinical data and its own algorithms can help to make the right choice. This trial is designed to assess the difference between retrospective electronic medical cards (EMC) therapy prescriptions and MedicBK prescriptions based on key patient characteristics.

DETAILED DESCRIPTION:
There is a lot of data from registries about poor adherence to guidelines. It is connected with a problem that patients usually have a lot of comorbidities and physicians need to know сonsequently the huge number of medications and combinations. It is very difficult to decide quickly according to available data from libraries like PubMed. The Clinical Decision Support Systems (CDSS) based on real clinical data and its own Artificial Intelligence algorithms can help to make the right choice. This trial is designed to assess the difference between retrospective electronic medical cards (EMC) therapy prescriptions and MedicBK prescriptions based on key patient characteristics.

Two groups of experts (cardiologists with clinical practice for more than 5 years) will be participating in the trial.

Using main characteristics from EMC the first group of experts will put this data into MedicBK platform and assess retrospective treatment. The next blinded group of experts will perform prescriptions using MedicBK algorithms based on current guidelines and data from available clinical trials. The main hypothesis is the use Clinical Decision Support Systems (CDSS) better than current clinical practice. This option can help to make the right choice of medical combination based on main patient's clinical characteristics

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patients diagnosed with nonvalvular atrial fibrillation and essential hypertension having indications for therapy according to European guidelines.

Exclusion Criteria:

1. Valvular cause of atrial fibrillation
2. GFR less than 30 ml / min
3. Active liver disease
4. Acute coronary syndrome
5. The presence of thyroid diseases as a cause of atrial fibrillation
6. Secondary arterial hypertension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with nonvalvular atrial fibrillation and essential hypertension having indications for therapy according to European guidelines
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Assessment of AF/AH treatment guidelines compliance | 1 MONTH
  Number of electronic medical records not compliant to the AF/AH clinical practice guidelines

SECONDARY OUTCOMES:
Assessment of MedicBK programme | 1 MONTH
  Number of prescriptions from electronic medical records appropriate or inappropriate according to the AF/hypertension clinical practice guidelines in comparison with the treatment's choice of CDSS platform

CONTACTS AND LOCATIONS:
Locations (1):
- V.A. Almazov Fnmrc, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No